CLINICAL TRIAL: NCT04174768
Title: The Effect of Bariatric Surgery on Glucose Metabolism and Kidney Function
Brief Title: The Effect of Bariatric Surgery on Glucose Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARDOM-Bari
Record Dates: First submitted 2019-11-17; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bariatric surgery patients (Experimental): Bariatric patients undergoing sleeve gastrectomy or Roux-en-Y gastric bypass
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery including sleeve gastrectomy and Roux-en-Y gastric bypass

SUMMARY:
This prospective, single arm, longitudinal study aims to assess the effect of bariatric surgery on glucose metabolism and kidney function.

DETAILED DESCRIPTION:
In recent years, it has become apparent that bariatric surgery not only promote dramatic weight loss but improve or eliminate type 2 diabetes (T2D). Furthermore, it has become increasingly clear that glucose homeostasis, which is mainly determined based on insulin secretion and insulin resistance, improves through mechanisms additional to the secondary consequences of weight reduction. We aims to assess the effect of bariatric surgery on glucose control and kidney function, and excavate potential mechanism for those effects.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years old
* body mass index ≥27.5 kg/m2, in case of type 2 diabetes
* body mass index ≥35 kg/m2, in case of non-type 2 diabetes

Exclusion Criteria:

* Prior complex gastrointestinal surgery, including that of the stomach, small intestine, large intestine, bile duct, pancreas, and spleen; Nissen, and trauma (except hemorrhoidectomy, herniorrhaphy, and appendectomy)
* Abdominal, thoracic, pelvic, and/or obstetric-gynecologic surgery within 3 months or at the discretion of the Investigator
* Cardiovascular conditions including significant known coronary artery disease (CAD), uncompensated congestive heart failure, history of stroke, or uncontrolled hypertension (defined as medially treated with the mean of three separate measurements systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg).

Subjects with CAD who were successfully treated with coronary artery bypass graft or percutaneous coronary intervention within 3 months and who have no evidence of active ischemia are eligible

* Kidney diseases including renovascular hypertension, renal artery stenosis, or end-stage renal disease
* Known history of chronic liver diseases including liver cirrhosis and alpha-1-antitrypsin deficiency
* Gastrointestinal disorders including a known history of celiac disease or any other malabsorptive disorders or inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Psychiatric disorders including dementia, active psychosis, history of suicide attempts, and alcohol or drug abuse within 12 months
* Severe pulmonary disease defined as forced expiratory volume at one second <50% of the predicted value
* Anemia defined as hemoglobin <8 in females and 10 in males
* Malignancy within 5 years (except squamous cell and basal cell cancer of the skin). Subjects diagnosed with early or stage 1 cancer that was successfully treated are eligible based on the Investigator's discretion
* Any condition or major illness that in the Investigator's judgement places the subject at undue risk by participating in the study
* Pregnancy
* Unable to understand the risks, realistic benefits, and compliance requirements of each program
* Use of investigational therapy or participation in any other clinical trial within 3 months
* Plans to move outside South Korea within the next 2 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-11-18 (Estimated); Study Completion 2021-11-18 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with diabetes remission | 12 months
  Remission (complete): Normal measures of glucose metabolism (HbA1c<6%, fasting plasma glucose<100mg/dl) in the absence antidiabetic medication

SECONDARY OUTCOMES:
Proportion of patients with optimal LDL cholesterol control | 3,6,12 months
  LDL cholesterol: <100 mg/dL = optimal (or <40 mg/dL if another risk factor is present)
Percent excess weight loss | 3,6,12 months
  Percent excess weight loss (%EWL) %EWL = [(Initial Weight) - (Postop Weight)]/[(Initial Weight) - (Ideal Weight)]
Changes of estimated glomerular filtration rate | 3,6,12 months
  Changes of Cystatin C or creatinine based eGFR Changes of urine protein(albumin) creatinine ratio
Changes of metabolites profile | 3,6,12 months
  Changes of serum diabetes-related metabolites profile including large neutral amino acids, tryptophan-derived metabolites
Proportion of patients with hypertension improvement | 3,6,12 months
  Improvement: Defined as a decrease in dosage or number of antihypertensive medication or decrease in systolic or diastolic blood pressure (BP) on the same medication (better control).

CONTACTS AND LOCATIONS:
Overall Officials: Sungsoo Park, MD,PhD, Principal Investigator — Korea University
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No